CLINICAL TRIAL: NCT05733156
Title: Abscopal Effect from the Addition of Low-dose Radiotherapy in Polymetastatic Cancer Patients Receiving Stereotactic Radiotherapy: a Multicenter, Single-arm Clinical Study (KROG 22-11)
Brief Title: Abscopal Effect from the Low-dose Radiotherapy in Polymetastatic Cancer Patients Receiving Stereotactic Radiotherapy
Acronym: KROG22-11
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Soonchunhyang University Hospital (Other)
Collaborators: SMG-SNU Boramae Medical Center (Other); Saint Vincent's Hospital, Korea (Other); Seoul National University Hospital (Other); Chungnam National University Hospital (Other)
Responsible Party: Principal Investigator, Ah Ram Chang, Director of Radiation Oncology, Soonchunhyang University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCHUH 2022-10-003
Record Dates: First submitted 2023-01-12; First posted 2023-02-17 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Neoplasms; Secondary Malignant Neoplasm
Keywords: Neoplasm Metastasis
MeSH Terms: conditions — Neoplasms; Neoplasms, Second Primary; Neoplasm Metastasis | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SBRT + LDRT (Experimental)
  Interventions: Radiation: SBRT + LDRT

INTERVENTIONS:
Radiation: SBRT + LDRT — Stereotactic body radiotherapy (SBRT) and low-dose radiotherapy (LDRT) are administered concurrently. SBRT is administered three times, at intervals of 1-2 days, and patients are treated with LDRT along with SBRT. LDRT is planned to irradiate EQD2 6 Gy considering the scattered dose caused by SBRT.

SUMMARY:
Recently, MD Anderson Cancer Center reported the phase II trial to investigate high-dose radiotherapy (HDRT, 20-70 Gy) and low-dose radiotherapy (LDRT, 1-10 Gy) for metastatic cancer patients who had undergone immunotherapy. HDRT or HDRT+LDRT was conducted in two respective groups and the treatment group was determined according to the disease status of participants, not randomization. Immunotherapy was maintained in this clinical study. Therefore, we aim to investigate this abscopal effect from adding LDRT to HDRT, irrespective of previous immunotherapy, in this multicenter, single-arm study.

ELIGIBILITY:
Inclusion Criteria:

* Patients who can provide their written informed consent
* Age ≥19 years
* Patients with histologically confirmed primary solid (irrespective of the status of the primary tumor)
* Patients with ECOG performance status 0-2
* Patients planning stereotactic body radiotherapy (three fractions) for extracranial metastases
* Based on RECIST v1.1, patients with at least one extracranial measurable lesion other than SBRT lesions
* Patients with one or more measurable lesions, which are not suitable for SBRT or palliative radiotherapy and can be considered for LDRT (bone metastasis is not indicated for LDRT)
* Patients with hematologic function suitable for radiotherapy (absolute neutrophil count ≥1,500/mm^3, hemoglobin ≥9 g/dL, platelet count ≥100,000/mm^3)
* Patients with a life expectancy of 6 months or more according to the researcher's judgment

Exclusion Criteria:

* Patients participating in other clinical studies that may affect the efficacy/safety of this clinical study
* Patients with brain metastasis
* Patients planning SBRT for all measurable lesions due to oligometastasis
* Patients with a history of radiotherapy for extracranial metastases within 3 months of the enrollment
* Patients unable to cooperate with stereotactic body radiotherapy
* Patients who are pregnant or planning to
* Patients with advanced or multiple malignancies requiring aggressive treatment (excluding skin cancers other than melanoma or intraepithelial cancer)
* Patients who have received systemic steroid therapy or immunosuppressive therapy within 2 weeks of enrollment - Patients with an (e.g. allergic disease, radiation pneumonitis, etc.) (The use of steroids for preventive purposes is allowed (e.g., to prevent vomiting during chemotherapy)) active autoimmune disease requiring systemic treatment within the past 2 years, evidence of clinically severe autoimmune disease, or syndrome requiring systemic steroid or immunosuppressive therapy (Patients who need intermittent use of bronchodilators, inhaled steroids, or topical steroid injections, hypothyroid patients on stable hormone replacement therapy, type 1 diabetes patients, or patients recovering from childhood asthma/atopic dermatitis are permitted)
* Patients with active infection requiring systemic treatment

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2023-01-03 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Abscopal effect rate of low-dose radiotherapy lesions | 3 months after completion of radiotherapy
  The proportion of patients with an abscopal response of low-dose radiotherapy lesions assessed by RECIST v1.1

SECONDARY OUTCOMES:
Abscopal effect rate of low-dose radiotherapy lesions | 1, 6, and 12 months after completion of radiotherapy
  The proportion of patients with an abscopal response of low-dose radiotherapy lesions assessed by RECIST v1.1
Overall response rate | 1, 3, 6, and 12 months after completion of radiotherapy
  The proportion of patients showing complete or partial response of metastatic lesions
Progression-free survival rate | 12 months after completion of radiotherapy
  From the date of enrollment to the date of progression or death assessed by RECIST v1.1
Overall survival rate | 12 months after completion of radiotherapy
  From the date of enrollment to the date of death or last follow-up assessed by RECIST v1.1
Adverse event | 12 months after completion of radiotherapy
  The proportion of patients with treatment-related adverse events as assessed by CTCAE v5.0
Immune cell subsets of peripheral blood and tissue samples | 1 and 3 months after completion of radiotherapy
  Number of immune cell count

CONTACTS AND LOCATIONS:
Overall Officials: Ah Ram Chang, MD, PhD, Study Chair — Soonchunhayng Universtiy Seoul Hospital
Locations (2):
- South Korea (2):
  - Seoul Metropolitan Government Seoul National University Boramae Medical Center, Seoul
  - Soonchunhyang University Seoul Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No